CLINICAL TRIAL: NCT02951767
Title: A Phase II, Multicenter, Single-Arm Study of Atezolizumab in Patients With Locally Advanced or Metastatic Urothelial Bladder Cancer
Brief Title: A Study of Atezolizumab in Participants With Locally Advanced or Metastatic Urothelial Bladder Cancer (Cohort 1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO29293 (Cohort 1); IMvigor 210 (Other: Genentech Inc.); 2013-005486-39 (EudraCT Number)
Expanded Access: NCT02589717 (Approved for marketing)
Record Dates: First submitted 2016-10-31; First posted 2016-11-01 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Bladder Cancer
Keywords: anti-PD-L1; PD-L1; MPDL3280A; PD-1; bladder cancer; atezolizumab; Tecentriq
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1: Treatment-naive Cisplatin Ineligible Participants (Experimental): Participants with advanced disease who are treatment-naive for advanced urothelial carcinoma and cisplatin ineligible will receive atezolizumab 1200 mg via IV infusion on Day 1 of 21-day cycles until disease progression per RECIST v1.1 criteria or unmanageable toxicity.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg will be given by IV infusion on Day 1 of 21-day cycles until disease progression per RECIST v1.1 criteria or unmanageable toxicity.
  Other Names: MPDL3280A; Tecentriq

SUMMARY:
This Phase II, single-arm study is designed to evaluate the effect of atezolizumab treatment in participants with locally advanced or metastatic urothelial bladder cancer. Participants will be enrolled into 1 of 2 cohorts. Cohort 1 (reported here) will consist of participants who are treatment-naïve and ineligible for cisplatin-containing chemotherapy. Cohort 2 will contain participants who have progressed during or following a prior platinum-based chemotherapy regimen. The results of the second cohort are reported separately (NCT02108652). Participants in both cohorts will be given a 1200 milligrams (mg) intravenous (IV) dose of atezolizumab on Day 1 of 21-day cycles. Treatment of participants in Cohort 1 will continue until disease progression per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) or unmanageable toxicity. Treatment of participants in Cohort 2 will continue until loss of clinical benefit or unmanageable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic transitional cell carcinoma of the urothelium (including renal pelvis, ureters, urinary bladder, urethra)
* Representative tumor specimens as specified by the protocol
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than or equal to (>=) 12 weeks
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end organ function

Cohort 1-Specific Inclusion Criteria

* No prior chemotherapy for inoperable locally advanced or metastatic or recurrent urothelial carcinoma
* Ineligible for cisplatin-based chemotherapy due to one of the following: Impaired renal function, a hearing loss of 25 decibels (dB) at two contiguous frequencies, Grade 2 or greater peripheral neuropathy, or ECOG performance score of 2

Exclusion Criteria:

* Any approved anti-cancer therapy within 3 weeks prior to initiation of study treatment
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrollment
* Active or untreated central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments
* Leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Uncontrolled hypercalcemia (greater than [>] 1.5 millimoles per liter [mmol/L] ionized calcium or Ca > 12 milligrams per deciliter [mg/dL] or corrected serum calcium > upper limits of normal [ULN]) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
* Malignancies other than urothelial bladder cancer within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome or incidental prostate cancer
* Pregnant and lactating women
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Serum albumin less than (<) 2.5 grams per deciliter (g/dL)
* Positive test for human immunodeficiency virus (HIV) and/or active hepatitis B or hepatitis C or tuberculosis
* Severe infections within 4 weeks prior to Cycle 1, Day 1
* Significant cardiovascular disease
* Major surgical procedure other than for diagnosis within 28 days prior to Cycle 1, Day 1
* Prior allogeneic stem cell or solid organ transplant
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4), anti-programmed death-1 receptor (anti-PD-1), and anti-programmed death-ligand 1 (anti-PD-L1) therapeutic antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-05-31 (Actual); Primary Completion 2016-07-04 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (77):
- United States (47):
  - University of Alabama At Birmingham, Birmingham, Alabama
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Arizona Oncology - HOPE Wilmot, Tucson, Arizona
  - UCLA, Los Angeles, California
  - The Angeles Clinic and Research Institute - W LA Office, Los Angeles, California
  - USC Norris Cancer Center, Los Angeles, California
  - UCSF, San Francisco, California
  - Kaiser Permanente - San Marcos, San Marcos, California
  - Stanford Cancer Center, Stanford, California
  - Kaiser Permanente; Oncology Clinical Trials, Vallejo, California
  - Rocky Mountain Cancer Center - Aurora, Aurora, Colorado
  - University Of Colorado, Aurora, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Yale Cancer Center ; Medical Oncology, New Haven, Connecticut
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - University of Chicago; Hematology/Oncology, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Indiana University Health; Goshen Center for Cancer Care, Goshen, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital;Oncology, Boston, Massachusetts
  - Dana Farber Cancer Inst. ; Dept. of Medical Oncology, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Harvard Medical School; Department of Medicine, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Urology Cancer Center & GU Research Network, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology, P.C., Albany, New York
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai School of Medicine - Tisch Cancer Institute, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Case Western Reserve Univ; Hem/Onc, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Willamette Valley Cancer Ctr - 520 Country Club, Eugene, Oregon
  - Kimmel Cancer Center Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Cancer Center - Tennessee Oncology, Pllc, Nashville, Tennessee
  - Ctr for Cancer and Blood Disorders, Fort Worth, Texas
  - Texas Oncology - Houston (Gessner), Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates - Lake Wright Cancer Center, Norfolk, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Canada (7):
  - Bcca - Cancer Center Southern Interior, Kelowna, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre; Oncology, Ottawa, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
- France (3):
  - APHP - Hospital Saint Louis, Paris
  - Hopital Foch; Oncologie, Suresnes
  - Institut Gustave Roussy; Oncologie Medicale, Villejuif
- Germany (5):
  - Charité - Universitätsmedizin Berlin; CC 8: Chirurgische Medizin; Klinik für Urologie, Berlin
  - Universitätsklinikum Düsseldorf; Urologische Klinik, Düsseldorf
  - Universitätsklinikum Freiburg; Chirurgische Klinik; Abteilung Urologie, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf Onkologisches Zentrum Medizinische Klinik II, Hamburg
  - Klinikum rechts der Isar der TU München; Urologische Klinik und Poliklinik, München
- Italy (2):
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Azienda USL8 Arezzo-Presidio Ospedaliero 1 San Donato;U.O.C. Oncologia, Arezzo, Tuscany
- The Netherlands Cancer Institute - Antoni Van Leeuwenhoekziekenhuis, Amsterdam, Netherlands
- Spain (7):
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
- United Kingdom (5):
  - University Hospital Birmingham The Cancer Centre, Queen Elizabeth Hospital, Birmingham
  - Barts and The London, London
  - Sarah Cannon Research Institute, London
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton

REFERENCES:
- [Derived] Szabados B, Ponz-Sarvise M, Machado R, Saldana D, Kadel EE, Banchereau R, Bouquet F, Garmhausen M, Powles T, Schroder C; imCORE Working Group of Early Career Investigators (imFLAME). Clinico-Genomic Characterization of Patients with Metastatic Urothelial Carcinoma in Real-World Practice Identifies a Novel Bladder Immune Performance Index (BIPI). Clin Cancer Res. 2022 Sep 15;28(18):4083-4091. doi: 10.1158/1078-0432.CCR-22-0200. PMID 35877091
- [Derived] Vander Velde N, Guerin A, Ionescu-Ittu R, Shi S, Wu EQ, Lin SW, Hsu LI, Saum KU, de Ducla S, Wang J, Li S, Thastrom A, Liu S, Shi L, Leppert JT. Comparative Effectiveness of Non-cisplatin First-line Therapies for Metastatic Urothelial Carcinoma: Phase 2 IMvigor210 Study Versus US Patients Treated in the Veterans Health Administration. Eur Urol Oncol. 2019 Feb;2(1):12-20. doi: 10.1016/j.euo.2018.07.003. Epub 2018 Aug 4. PMID 30929841

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is considered "Completed" because the planned study activities and analyses have been performed.
Pre-assignment Details: The analysis included data up to cutoff date 28 February 2023.
Groups:
- Cohort 1: Treatment-naive Cisplatin Ineligible Participants: Participants with advanced disease who were treatment-naive for advanced urothelial carcinoma and cisplatin ineligible received atezolizumab 1200 milligrams (mg) via intravenous (IV) on Day 1 of 21-day cycles until disease progression per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) criteria or unmanageable toxicity.
Period: Overall Study
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Started | 119
Completed | 0
Not Completed | 119
Not completed — Study Terminated By Sponsor | 9
Not completed — Withdrawal by Subject | 11
Not completed — Death | 96
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Cohort 1 Safety Evaluable Population included all participants who received any amount of study drug.
Groups:
- Cohort 1: Treatment-naive Cisplatin Ineligible Participants: Participants with advanced disease who were treatment-naive for advanced urothelial carcinoma and cisplatin ineligible received atezolizumab 1200 mg via IV infusion on Day 1 of 21-day cycles until disease progression per RECIST v1.1 criteria or unmanageable toxicity.
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Confirmed Objective Response of Complete Response (CR) or Partial Response (PR) as Assessed by the Independent Review Facility (IRF) According to RECIST v1.1
Description: Tumor response was assessed by the IRF according to RECIST v1.1. CR was defined as disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as greater than or equal to (≥) 30 percent (%) decrease in sum of longest diameter (LD) of target lesions in reference to Baseline sum LD. Response was to be confirmed ≥4 weeks after the initial assessment of CR or PR. The percentage of participants with a confirmed objective response of CR or PR was reported. The exact 95% confidence interval (CI) was calculated using the Clopper-Pearson method.
Time Frame: Baseline until confirmed disease progression or death, whichever occurred first (assessed at every 9 weeks for the first 12 months, thereafter every 12 weeks until data cutoff date 04 July 2016, up to maximum length of follow-up of 23.52 months)
Population: Cohort 1 objective response-evaluable population included intent-to-treat (ITT) participants who had measurable disease per RECIST v1.1 at baseline. Cohort 1 ITT population included all participants from Cohort 1 who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 119
percentage of participants | 22.7 [15.5 to 31.3]

2. Secondary Outcome: Duration of Response (DOR) as Assessed by the IRF According to RECIST v1.1
Description: DOR was defined as the time from the initial occurrence of documented CR or PR (whichever occurred first) until documented disease progression or death due to any cause on study, whichever occurred first. Tumor response was assessed by the IRF according to RECIST v1.1. CR was defined as disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in sum of LD of target lesions in reference to Baseline sum LD. Response was to be confirmed ≥4 weeks after the initial assessment of CR or PR.
Time Frame: as for outcome 1
Population: Cohort 1 objective response-evaluable population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 27
months | NA [3.7 to NA] — The median DOR and upper limit for the Full Range were not reached at a median follow up of 17.216 months on study.

3. Secondary Outcome: DOR as Assessed by the Investigator According to RECIST v1.1
Description: DOR was defined as the time from the initial occurrence of documented CR or PR (whichever occurred first) until documented disease progression or death due to any cause on study, whichever occurred first. Tumor response was assessed by the investigator according to RECIST v1.1. CR was defined as disappearance of all target and non-target lesions and no new measurable or unmeasurable lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in sum of LD of target lesions in reference to Baseline sum LD.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 30
months | NA [4.3 to NA] — The median DOR and upper limit for the Full Range were not reached at a median follow up of 17.216 months on study.

4. Secondary Outcome: Percentage of Participants With Death or Disease Progression as Assessed by the IRF According to RECIST v1.1
Description: Tumor response was assessed by the IRF according to RECIST v1.1. Disease progression or PD was defined as ≥20% increase in sum LD in reference to the smallest on-study sum LD, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: Cohort 1 ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 119
percentage of participants | 73.9 [2 to NA]

5. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by the IRF According to RECIST v1.1
Description: PFS was defined as the time from start of treatment to the first event of death or PD. Tumor response was assessed by the IRF according to RECIST v1.1. Disease progression or PD was defined as ≥20% increase in sum LD in reference to the smallest on-study sum LD, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: Cohort 1 ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 119
months | 2.69 [2.10 to 4.17]

6. Secondary Outcome: Percentage of Participants With Death or Disease Progression as Assessed by the Investigator According to RECIST v1.1
Description: Tumor response was assessed by the investigator according to RECIST v1.1. Disease progression or PD was defined as ≥20% increase in sum LD in reference to the smallest on-study sum LD, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The percentage of participants who died or experienced PD was reported.
Time Frame: as for outcome 1
Population: Cohort 1 ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 119
percentage of participants | 71.4 [2 to NA]

7. Secondary Outcome: PFS as Assessed by the Investigator According to RECIST v1.1
Description: PFS was defined as the time from start of treatment to the first event of death or PD. Tumor response was assessed by the investigator according to RECIST v1.1. Disease progression or PD was defined as ≥20% increase in sum LD in reference to the smallest on-study sum LD, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: Cohort 1 ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 119
months | 4.17 [2.3 to 5.75]

8. Secondary Outcome: Percentage of Participants With a Confirmed Objective Response of CR or PR as Assessed by the Investigator According RECIST v1.1
Description: Tumor response was assessed by the investigator according to RECIST v1.1. CR was defined as disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in sum of LD of target lesions in reference to Baseline sum LD. Response was to be confirmed ≥4 weeks after the initial assessment of CR or PR. The percentage of participants with a confirmed objective response of CR or PR was reported. The exact 95% CI was calculated using the Clopper-Pearson method.
Time Frame: as for outcome 1
Population: Cohort 1 objective response-evaluable population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 119
percentage of participants | 25.2 [17.7 to 34.0]

9. Secondary Outcome: Percentage of Participants Who Died
Description: The percentage of participants who died from any cause was reported.
Time Frame: Baseline until death (data cutoff date 04 July 2016, up to maximum length of follow-up of 23.52 months)
Population: Cohort 1 ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 119
percentage of participants | 49.6 [15.52 to 31.27]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from start of treatment to the time of death from any cause on study.
Time Frame: Baseline until death (data cutoff date 04 July 2016, up to maximum length of follow-up of 23.52 months)
Population: Cohort 1 ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 119
months | 15.9 [10.4 to NA] — The upper limit of the 95% CI was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

11. Secondary Outcome: Percentage of Participants Alive at 1-year
Time Frame: 1-year
Population: Cohort 1 ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 119
percentage of participants | 57.2 [48.2 to 66.3]

12. Secondary Outcome: Maximum Serum Concentration (Cmax) of Atezolizumab
Time Frame: Pre-dose (0 hours) and 30 minutes post-dose on Day 1 of Cycle 1 (Cycle length = 21 days)
Population: Cohort 1 pharmacokinetic (PK) evaluable population was defined as participants who received any dose of atezolizumab treatment and had PK data at timepoints that were sufficient to determine PK parameters. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: microgram(s)/milliliter (mcg/mL)
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 113
microgram(s)/milliliter (mcg/mL) | 386 (118) [36.29 to 62.3]

13. Secondary Outcome: Minimum Serum Concentration (Cmin) of Atezolizumab
Time Frame: Pre-dose (0 hours) on Day 1 of Cycles 1, 2, 3, 4, 8 (Cycle length = 21 days)
Population: Cohort 1 PK evaluable population. Here, number of participants analyzed = participants who were evaluable for this outcome. "n" = participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 117
mcg/mL
  Pre-dose Cycle 1 (n=117) | 0 (0) [36.29 to 62.3]
  Pre-dose Cycle 2 (n=106) | 77.7 (35.3)
  Pre-dose Cycle 3 (n=57) | 117 (48.8)
  Pre-dose Cycle 4 (n=66) | 159 (68.4)
  Pre-dose Cycle 8 (n=47) | 169 (110)

14. Secondary Outcome: Percentage of Participants Positive for Anti-therapeutic Antibodies (ATA) to Atezolizumab
Time Frame: Day 1 of all cycles (Cycle length = 21 days) and at treatment discontinuation (data cutoff date 04 July 2016, up to maximum length of follow-up of 23.52 months)
Population: Cohort 1 Safety Evaluable Population. Here, number of participants analyzed = participants for whom ATA samples were available.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Treatment-naive Cisplatin Ineligible Participants
Number analyzed (Participants) | 111
percentage of participants | 47.7 (0) [36.29 to 62.3]

ADVERSE EVENTS:
Time Frame: First dose of study drug until data cutoff date 28 February 2023 (up to approximately 105 months)
Description: All-Cause Mortality was assessed for all enrolled participants, Serious and Other Adverse Events were assessed in the safety population.
Arm/Group | MPDL3280A COHORT1 INFUSION
All-Cause Mortality (participants affected / at risk) | 96/119
Serious Adverse Events (participants affected / at risk) | 49/119
Other Adverse Events (participants affected / at risk) | 110/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPDL3280A COHORT1 INFUSION (N=119)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1)
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 (0)
AUTOIMMUNE COLITIS (Gastrointestinal disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 2 (2)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (5)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 (3)
SUBILEUS (Gastrointestinal disorders) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1)
ASTHENIA (General disorders) | 2 (2)
CHILLS (General disorders) | 0 (0)
FATIGUE (General disorders) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0)
HAEMORRHAGIC CYST (General disorders) | 0 (0)
MALAISE (General disorders) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
PAIN (General disorders) | 0 (0)
PERFORMANCE STATUS DECREASED (General disorders) | 0 (0)
PYREXIA (General disorders) | 1 (1)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1)
ABDOMINAL INFECTION (Infections and infestations) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1)
BILIARY SEPSIS (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0)
BURSITIS INFECTIVE STAPHYLOCOCCAL (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
CELLULITIS OF MALE EXTERNAL GENITAL ORGAN (Infections and infestations) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 0 (0)
MENINGOENCEPHALITIS HERPETIC (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2)
POST PROCEDURAL INFECTION (Infections and infestations) | 1 (1)
PULMONARY SEPSIS (Infections and infestations) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0)
RETROPERITONEAL INFECTION (Infections and infestations) | 0 (0)
SEPSIS (Infections and infestations) | 3 (3)
SKIN INFECTION (Infections and infestations) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 4 (4)
URINARY TRACT INFECTION PSEUDOMONAL (Infections and infestations) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0)
ILIUM FRACTURE (Injury, poisoning and procedural complications) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0)
STOMA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0)
VASCULAR PSEUDOANEURYSM RUPTURED (Injury, poisoning and procedural complications) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0)
TUMOUR ASSOCIATED FEVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0)
ATAXIA (Nervous system disorders) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0)
DIPLEGIA (Nervous system disorders) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0)
PARAPLEGIA (Nervous system disorders) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (2)
THROMBOSIS IN DEVICE (Product Issues) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 4 (5)
BLADDER PERFORATION (Renal and urinary disorders) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0)
HYDROURETER (Renal and urinary disorders) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 3 (3)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0)
PENILE PAIN (Reproductive system and breast disorders) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0)
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DERMATITIS PSORIASIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0)
IMMOBILE (Social circumstances) | 0 (0)
RENAL STONE REMOVAL (Surgical and medical procedures) | 0 (0)
URETERAL STENT INSERTION (Surgical and medical procedures) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
EMBOLISM (Vascular disorders) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPDL3280A COHORT1 INFUSION (N=119)
ANAEMIA (Blood and lymphatic system disorders) | 25 (39)
HYPOTHYROIDISM (Endocrine disorders) | 10 (10)
ABDOMINAL PAIN (Gastrointestinal disorders) | 14 (15)
CONSTIPATION (Gastrointestinal disorders) | 21 (35)
DIARRHOEA (Gastrointestinal disorders) | 31 (50)
NAUSEA (Gastrointestinal disorders) | 29 (35)
VOMITING (Gastrointestinal disorders) | 24 (29)
ASTHENIA (General disorders) | 12 (18)
CHILLS (General disorders) | 11 (16)
FATIGUE (General disorders) | 64 (87)
OEDEMA PERIPHERAL (General disorders) | 23 (30)
PAIN (General disorders) | 7 (8)
PYREXIA (General disorders) | 21 (24)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (13)
URINARY TRACT INFECTION (Infections and infestations) | 21 (30)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 10 (17)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 10 (26)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 8 (12)
BLOOD CREATININE INCREASED (Investigations) | 22 (35)
LYMPHOCYTE COUNT DECREASED (Investigations) | 7 (13)
WEIGHT DECREASED (Investigations) | 12 (13)
DECREASED APPETITE (Metabolism and nutrition disorders) | 37 (46)
DEHYDRATION (Metabolism and nutrition disorders) | 10 (10)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 11 (21)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 11 (19)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 12 (26)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 27 (45)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 19 (21)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 6 (6)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 6 (7)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 (17)
DIZZINESS (Nervous system disorders) | 10 (13)
HEADACHE (Nervous system disorders) | 13 (17)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 6 (6)
ANXIETY (Psychiatric disorders) | 11 (12)
CONFUSIONAL STATE (Psychiatric disorders) | 7 (10)
DEPRESSION (Psychiatric disorders) | 7 (7)
INSOMNIA (Psychiatric disorders) | 12 (12)
DYSURIA (Renal and urinary disorders) | 6 (6)
HAEMATURIA (Renal and urinary disorders) | 12 (15)
PROTEINURIA (Renal and urinary disorders) | 6 (8)
PELVIC PAIN (Reproductive system and breast disorders) | 7 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 25 (29)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 18 (18)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 7 (8)
DRY SKIN (Skin and subcutaneous tissue disorders) | 10 (10)
PRURITUS (Skin and subcutaneous tissue disorders) | 23 (39)
RASH (Skin and subcutaneous tissue disorders) | 14 (22)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 6 (6)
HYPOTENSION (Vascular disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.